CLINICAL TRIAL: NCT02670616
Title: Phase II Study of Ibrutinib in Combination With Rituximab-CHOP in Epstein-Barr Virus-positive Diffuse Large B-cell Lymphoma 54179060LYM2003 (Nick Name: IVORY Study)
Brief Title: Study of Ibrutinib in Combination With Rituximab-CHOP in Epstein-Barr Virus-positive Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-04-027
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Epstein-Barr Virus-positive Diffuse Large B-cell Lymphoma
MeSH Terms: interventions — ibrutinib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ibrutinib in combination with r-CHOP (Experimental): Ibrutinib560 mg daily on day 1-21 per each cycle ,Rituximab375 mg/m2, Cyclophosphamide750 mg/m2, doxorubicin 50 mg/m2, vincristine1.4 mg/m2 on day 1; Prednisolone 100mg per day on day 1-5 ,cycle length: 21 days ,Six cycles of treatment
  Interventions: Drug: Ibrutinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: vincristine; Drug: Prednisolone

INTERVENTIONS:
Drug: Ibrutinib — 560 mg by mouth daily on day 1-21 per each cycle
  Other Names: Imbruvica
Drug: Rituximab — 375 mg/m2 IV, day 1
  Other Names: Mabthera
Drug: Cyclophosphamide — 750 mg/m2 IV day 1
  Other Names: Endoxan
Drug: Doxorubicin — 50 mg/m2 IV day 1
  Other Names: Adriamycin
Drug: vincristine — 1.4 mg/m2 IV on day 1
Drug: Prednisolone — 100mg per day on day 1-5
  Other Names: solondo

SUMMARY:
This study was conducted to evaluate the complete response rate of Ibrutinib + R-CHOP in patients with Epstein-Barr virus-positive diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
EBV-positive diffuse large B-cell lymphoma has EBV-mediated carcinogenic signaling pathway activation, and this diverse intracellular pathway may be a potential therapeutic target in this disease.

The BTK inhibitor, ibrutinib, targets the B cell receptor signaling pathway and is active against B cell non-Hodgkin lymphoma. As a result, evidence of the antitumor effect of ibrutinib has been accumulated in some B-cell lymphoma forms such as mantle cell lymphoma. The addition of ibrutinib to standard chemotherapy, rituximab-CHOP, is considered to be an effective treatment for patients with EBV-positive diffuse large B-cell lymphomas, because it is known to show a poor response to treatment compared to (NOS) diffuse large B- It can provide benefits to patients.

The BTK inhibitor, ibrutinib, targets the B cell receptor signaling pathway and is active against B cell non-Hodgkin lymphoma. As a result, evidence of the antitumor effect of ibrutinib has been accumulated in some B-cell lymphoma forms such as mantle cell lymphoma. The addition of ibrutinib to standard chemotherapy, rituximab-CHOP, is considered to be an effective treatment for patients with EBV-positive diffuse large B-cell lymphomas, because it is known to show a poor response to treatment compared to (NOS) diffuse large B- It can provide benefits to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, histologically proven EBV-positive Diffuse large B-cell lymphoma A.EBV positivity: The presence of EBER-positive tumor cells ≥ 20% B.DLBCL based on the WHO classification 2008
2. Hematology values must be within the following limits:

   A.Absolute neutrophil count 1000/mm3 independent of growth factor support B.Platelets 100,000/mm3 or 50,000/mm3 if bone marrow involvement independent of transfusion support in either situation C.Hemoglobin ≥ 10.0 g/dL (may be transfused or erythropoietin treated)
3. Biochemical values within the following limits:

   A.Alanine aminotransferase and aspartate aminotransferase≤ 3 x upper limit of normal B.Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin C.Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft Gault) ≥ 40 mL/min/1.73m2 D.Serum calcium ≤ 12.0 mg/dL
4. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug
5. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin)or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
6. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.
7. At least one measurable lesion
8. ECOG PS 0-2
9. Informed consent
10. Age ≥ 19 years

Exclusion Criteria:

1. Previous treatment history for EBV-positive DLBCL including any kinds of chemotherapy

   •Exception: a) Prednisolone 100mg or equivalent dosage of any types of steroid is allowed (Maximum 7 days); b) Radiation for reducing symptom related with mass effect is allowed
2. History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease or secondary CNS involvement on CT or MRI scan.
3. Pregnancy or breastfeeding
4. Major surgery within 4 weeks of enrollment
5. History of stroke or intracranial hemorrhage within 6 months prior to enrollment
6. Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon).
7. Requires treatment with strong CYP3A inhibitors.
8. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
9. Vaccinated with live, attenuated vaccines within 4 weeks of enrollment.
10. Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
11. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
complete response rate | From date of enrollment until the date first documented disease progression or unacceptable toxicity, whichever came first, assessed up to 48 months
  To assess the efficacy of disease control including complete response (CR), partial response (PR) and stable disease (SD)

SECONDARY OUTCOMES:
Progression-free survival | the time between the date of treatment start and the date of death due to any cause or date of disease progression..assessed up to 48 months
  It is a measure of the period of survival without disease progression
Overall survival (OS) | Time between the start of treatment and the date of death.assessed up to 48 months
  It measures the time from start of treatment to death.
Toxicity Profile | from the date of informed consent signature to 30 days after last drug administration.
  Clinical and laboratory toxicity/symptomatology will be graded based on the NCIC CTG v4.03. Adverse events not reported in NCIC CTG will be categorized into mild, moderate, severe, and fatal and further classified to CTCAE Grades 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Won seog KIM, MD,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Gangnam-gu, South Korea